CLINICAL TRIAL: NCT05924893
Title: The Use of Naltrexone Hydrochloride to Promote Healing in Patients With Resistant Non-infectious Corneal Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahemd Abdelghany, Associate professor, Minia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015
Record Dates: First submitted 2023-06-11; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Cornea Ulcer
MeSH Terms: conditions — Corneal Ulcer | interventions — Naltrexone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naltrexone group (Experimental): 25 eyes with refractory non infective corneal ulcer were subjected to daily insertion of a NTX film in the lower conjunctival fornix for 2 weeks
  Interventions: Drug: Naltrexone Hydrochloride
- Control (Experimental): 25 eyes with refractory non infective corneal ulcer were treated by carboxymethyl cellulose sodium 0.5 % eye drops
  Interventions: Drug: Carboxy methyl cellulose

INTERVENTIONS:
Drug: Naltrexone Hydrochloride — naltrexone film
  Other Names: NTX
  Arms: Naltrexone group
Drug: Carboxy methyl cellulose — Carboxy methyl cellulose drops
  Other Names: Carboxy methyl cellulose sodium 0.5%
  Arms: Control

SUMMARY:
The opioid growth factor-receptor antagonist-naltrexone hydrochloride (NTX)- has gained much reach interest for applications in ophthalmology, because of its novel mechanism of action for speeding up corneal wound healing in both diabetics and non-diabetics, effective both locally and systemically and its availability as a low molecular weight synthetic drug.

DETAILED DESCRIPTION:
Corneal epithelial defects generally heal within 2 days without complications, in some patients with decreased corneal sensitivity, such as patients with severe dry eye, corneal neuropathy, or autoimmune diseases, the corneal epithelium shows a reduced tendency for spontaneous healing Resistant corneal ulcers may appear as epithelial defects associated to Bowman's layer disruption with associated damage and partial variable loss of superficial corneal stroma larger than 2 mm in diameter that persist more than 2 weeks even treated with conventional treatment . Noninfectious corneal ulcers have a similar clinical presentation like that of infectious ulcers but with no known infectious cause . Resistant corneal ulcer can lead to serious complications such as infection, inflammation, corneal scarring, opacification, corneal thinning, and perforation . In our study NTX accelerated healing of resistant corneal ulcers that was refractory to conventional treatment with lubricant eye drops and was safe with no complications reported in all treated eyes.

ELIGIBILITY:
Inclusion Criteria:

* refractory non infective corneal ulcer

Exclusion Criteria:

* infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
healing of ulcer | 2 weeks
  healing of ulcer measured in millemeters by clinical examination on slit lamp after staining with sodium fluorescein stain

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Moharram, professor, Principal Investigator — Minia University
Locations (1):
- Faculty of Medicine, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alio JL, Abad M, Artola A, Rodriguez-Prats JL, Pastor S, Ruiz-Colecha J. Use of autologous platelet-rich plasma in the treatment of dormant corneal ulcers. Ophthalmology. 2007 Jul;114(7):1286-1293.e1. doi: 10.1016/j.ophtha.2006.10.044. Epub 2007 Feb 26. PMID 17324465